CLINICAL TRIAL: NCT06003946
Title: Effectiveness of a Breathing and Relaxation Technique in Antenatal Education (BreLax Study): a Randomised Controlled Trial
Brief Title: Effectiveness of a Breathing and Relaxation Technique in Antenatal Education
Acronym: BreLax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Principal Investigator, Vanessa Leutenegger, PhD Student, Zurich University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023 - 000183124; ZHAW (Other: Zurich University of Applied Sciences); UZH (Other: University of Zurich)
Record Dates: First submitted 2023-07-27; First posted 2023-08-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: breathing technique; birth preparation; prenatal education
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (BreLax) (Experimental): BreLax: midwife-led antenatal education class
  Interventions: Behavioral: BreLax: Antenatal education class
- Control group (Standard care) (Active Comparator): Midwife-led antenatal education class
  Interventions: Behavioral: Standard care (control)

INTERVENTIONS:
Behavioral: BreLax: Antenatal education class — An antenatal education class over 9 hours with information regarding pregnancy, labour and birth, pain management as well as the postpartum period with an integrated breathing and relaxation technique (prolonged exhalation in the individual rhythm) and 4 accompanying positions (standing upright, sitting supported, four-footed, supported lying on the side). In addition, participants receive a manual for independent practice at home.
  Arms: Intervention group (BreLax)
Behavioral: Standard care (control) — An antenatal education class over 9 hours, with information regarding pregnancy, labour and birth, pain management and the postpartum period as well as some relaxation exercises.
  Arms: Control group (Standard care)

SUMMARY:
The aim of this randomised controlled trial is to compare the effects of an antenatal education class including a breathing and relaxation technique on self-efficacy compared to a standard antenatal education class without a focus on breathing and relaxation techniques.

DETAILED DESCRIPTION:
Antenatal education classes were developed to inform expectant mothers about pregnancy, labour and birth and the postpartum period with the aim of improving pregnancy and childbirth experience. They were based, for example, on concepts of Lamaze and Grantly Dick-Read. Studies indicate positive emotional effects on labour and birth outcomes in women who attended antenatal education classes. This includes lower levels of fear of childbirth, lower rates of caesarean birth at the women's request, a higher rate of spontaneous births, and a stronger involvement of the partner, better chances of initiating breastfeeding, a lower likelihood of developing depression symptoms during the postpartum period. There is limited evidence on the link between birth preparation and neonatal outcomes. Considering recent evidence suggesting that antenatal education classes may positively influence maternal and neonatal birth outcomes, we intend to analyse an antenatal education class focusing on a breathing and relaxation technique and assess the impact of such a class on self-efficacy, as well as other maternal and neonatal birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a singleton low-risk pregnancy
* receiving antenatal care
* being willing to attend an antenatal education class
* planning a vaginal birth
* sufficient oral and written German language knowledge

Exclusion Criteria:

* women, who plan an elective caesarean section
* pregnant with multiples
* do not have sufficient oral and written German language knowledge

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 13 weeks till 37 weeks of pregnancy
  Changes from baseline to after the antenatal education class measured with the german version of the childbirth self-efficacy inventory (CBSEI).
  The CBSEI is a 32-item scale that measures women's perceived self-efficacy towards labour. Items are scored on a scale of 1 to 10. A higher score indicates that participants are better able to cope with difficult tasks.

SECONDARY OUTCOMES:
Childbirth experience | within 4 weeks after birth
  Birth experience is assessed after birth using the german version of the childbirth experience questionnaire (CEQ 2.0) The CEQ 2.0 is a 25-item scale with four dimensions (own capacity, perceived safety, professional support and participation). Items are scored on a scale of 1 (disagree at all) to 4 (agree completely). A higher value indicates a more positive assessment of the birth experience.
pain management | within 4 weeks after birth
  epidural anesthesia (PDA) yes/no, nitrous oxide yes/no, Patient Controlled Analgesia (PCA) yes/no, other pain medication yes/no (medical birth record)
birthing position | within 4 weeks after birth
  Documented during labour and birth (medical birth record). elevated supine yes/no, lateral position yes/no, standing yes/no, 4-foot position yes/no, bathtub yes/no, sitting (stool) yes/no
Duration of labour | within 4 weeks after birth
  Documented during labour and birth (medical birth record)
Bonding | within 4 weeks after birth
  Documented during labour and birth (medical birth record). Direct skin contact after birth (Bonding) yes/no
5-minute Apgar-Score | within 4 weeks after birth
  Documented during labour and birth (medical birth record). Appearance 0 to 2 (pale/ trunk rosy, extremities pale/ rosy), Pulse 0 to 2 (no Puls/ <100/min/ >100/min), Grimace 0 to 2 (No/ Grimacing/ Screaming), Activity 0 to 2 (Flaccid/ Sluggish flexion movements/ Spontaneous good self-movement), Respiration 0 to 2 (None/ Slow, irregular breathing or gasping/ Regular (40/min)). Interpretation: normal: 9-10 points; marginal: 5-8 points; critical for the newborn: <5 points.
arterial umbilical cord pH | within 4 weeks after birth
  Documented after labour and birth (medical birth record). Normal values in the umbilical artery blood are values of 7.20 - 7.38. At pH below 7.2 there is mild acidosis, below 7.1 moderate acidosis and below 7.0 severe acidosis.
Feasibility and effectiveness BreLax | 13 weeks of pregnancy till 4 weeks after birth
  Self-reported by participants (digital diary and questionnaire). How often practiced before birth (text), how long practiced each time (Text) , where practiced (Text) , when used during birth (contractions irregular yes/no, contractions regular yes/no, at end of birth (pushing phase) yes/no, whole birth) yes/no.

CONTACTS AND LOCATIONS:
Locations (1):
- Zurich University of Applied Sciences, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shand AW, Lewis-Jones B, Nielsen T, Svensson J, Lainchbury A, Henry A, Nassar N. Birth outcomes by type of attendance at antenatal education: An observational study. Aust N Z J Obstet Gynaecol. 2022 Dec;62(6):859-867. doi: 10.1111/ajo.13541. Epub 2022 May 17. PMID 35581951
- [Background] Rouhe H, Salmela-Aro K, Toivanen R, Tokola M, Halmesmaki E, Saisto T. Obstetric outcome after intervention for severe fear of childbirth in nulliparous women - randomised trial. BJOG. 2013 Jan;120(1):75-84. doi: 10.1111/1471-0528.12011. Epub 2012 Nov 2. PMID 23121002
- [Background] Svensson J, Barclay L, Cooke M. Randomised-controlled trial of two antenatal education programmes. Midwifery. 2009 Apr;25(2):114-25. doi: 10.1016/j.midw.2006.12.012. Epub 2007 Apr 24. PMID 17459542
- [Background] Svensson J, Barclay L, Cooke M. Effective antenatal education: strategies recommended by expectant and new parents. J Perinat Educ. 2008 Fall;17(4):33-42. doi: 10.1624/105812408X364152. PMID 19436529
- [Background] Ip WY, Tang CS, Goggins WB. An educational intervention to improve women's ability to cope with childbirth. J Clin Nurs. 2009 Aug;18(15):2125-35. doi: 10.1111/j.1365-2702.2008.02720.x. PMID 19583645
- [Background] Ahlden I, Ahlehagen S, Dahlgren LO, Josefsson A. Parents' expectations about participating in antenatal parenthood education classes. J Perinat Educ. 2012 Winter;21(1):11-7. doi: 10.1891/1058-1243.21.1.11. PMID 23277726
- [Background] Schmidt G, Stoll K, Jager B, Gross MM. [German Version of the Childbirth Self-Efficacy Inventory and its Short Form]. Z Geburtshilfe Neonatol. 2016 Feb;220(1):28-34. doi: 10.1055/s-0035-1547296. Epub 2015 Sep 17. German. PMID 26378776
- [Derived] Leutenegger V, Wieber F, Daly D, Sultan-Beyer L, Bagehorn J, Pehlke-Milde J. Study protocol of a breathing and relaxation intervention included in antenatal education: A randomised controlled trial (BreLax study). PLoS One. 2024 Oct 8;19(10):e0308480. doi: 10.1371/journal.pone.0308480. eCollection 2024. PMID 39378237

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT06003946/Prot_SAP_000.pdf